CLINICAL TRIAL: NCT06970964
Title: A Multi-Center, Double-Blind, Randomized, Parallel Group Study to Evaluate the Effect of Fermented Milk Containing Lacticaseibacillus Paracasei Strain Shirota (LCS) on the Upper Airway Symptoms of Triathletes Both Before and After a Competition
Brief Title: Fermented Milk Drink With Lacticaseibacillus Paracasei Strain Shirota Helps Triathletes With Cold-Like Symptoms Before and After a Race
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Jonatas Bussador do Amaral, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 7.349.261
Record Dates: First submitted 2025-04-30; First posted 2025-05-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Tract Infections (RTI); Mucosal Immunity; Systemic Inflammation; Depressive Disorder; Exercise-Induced Immunosuppression; Athletic Performance; Upper Respiratory Tract Symptoms; Mental Health; Cytokine Response; Probiotic Therapy
Keywords: Immune Function; Sports Nutrition; Endurance Athletes; Lacticaseibacillus paracasei strain Shirota; Upper Respiratory Symptoms; Respiratory Tract Infections; Immunity; Mucosal; Inflammation; Probiotics; Exercise
MeSH Terms: conditions — Respiratory Tract Infections; Depressive Disorder; Psychological Well-Being; Signs and Symptoms, Respiratory; Inflammation; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: one receiving fermented milk containing Lacticaseibacillus paracasei strain Shirota and the other receiving placebo (non-fermented milk).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Participants, care providers, investigators, and outcomes assessors will be blinded to group assignments to prevent bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Participants will receive one bottle per day of fermented milk containing 40 billion colony-forming units of Lacticaseibacillus paracasei strain Shirota (LcS) for 44 days.Intervention:
  Type: Dietary Supplement Name: Lacticaseibacillus paracasei strain Shirota Description: Daily intake of fermented milk containing 40 billion CFU of LcS.
  Interventions: Dietary Supplement: Intervention Name: Fermented milk containing Lacticaseibacillus paracasei strain Shirota. Intervention Name: Non-fermented milk (placebo)
- Placebo Group (Placebo Comparator): Name: Non-fermented milk Description: Daily intake of placebo (non-fermented milk) matched in appearance and taste to the probiotic.
  Interventions: Dietary Supplement: Non-fermented milk (placebo)

INTERVENTIONS:
Dietary Supplement: Intervention Name: Fermented milk containing Lacticaseibacillus paracasei strain Shirota. Intervention Name: Non-fermented milk (placebo) — Participants will ingest 80 mL per day of fermented milk containing 40 billion colony-forming units (CFU) of Lacticaseibacillus paracasei strain Shirota (LcS), starting 30 days before a triathlon competition and continuing until 14 days post-race. The fermented milk is stored refrigerated and consumed once daily.
  Other Names: LcS; Lacticaseibacillus casei Shirota; Probiotic milk drink
  Arms: Probiotic
Dietary Supplement: Non-fermented milk (placebo) — Participants will ingest 80 mL per day of non-fermented milk identical in taste, appearance, and packaging to the probiotic drink, but without Lacticaseibacillus paracasei strain Shirota. Administration follows the same schedule as the probiotic group.
  Other Names: Placebo milk
  Arms: Placebo Group

SUMMARY:
This study aims to evaluate whether a fermented milk drink containing the probiotic strain Lacticaseibacillus paracasei strain Shirota (LCS), commonly found in Yakult®, can help reduce upper respiratory symptoms in triathletes before and after competition.

Athletes often experience cold-like symptoms due to physical stress, intense training, and immune system challenges. The study investigates whether daily consumption of this probiotic drink can help improve immune response and reduce the incidence or severity of symptoms such as sore throat, nasal congestion, or coughing.

This is a randomized, double-blind, placebo-controlled, parallel-group study involving healthy adult triathletes. Participants will be randomly assigned to receive either the probiotic drink or a placebo for a specific period before and after a triathlon event. Symptoms and health markers will be tracked through questionnaires and biological samples.

The goal is to explore whether probiotic supplementation can provide practical, non-pharmacological support for athletes' immune health and well-being during intense physical activity.

DETAILED DESCRIPTION:
Background:

Endurance athletes are frequently exposed to high physical stress, which may lead to temporary immune suppression and increased susceptibility to upper respiratory tract infections (URTIs). Previous studies suggest that probiotics may play a role in supporting the immune system.

Objective:

To assess the efficacy of a fermented milk drink containing Lacticaseibacillus paracasei strain Shirota (LCS) in reducing upper airway symptoms in triathletes before and after a competitive event.

Study Design:

This is a multi-center, double-blind, randomized, placebo-controlled, parallel-group study. Eligible participants will be healthy adult triathletes preparing for a scheduled race. They will be randomized to consume either the probiotic drink or a placebo daily, starting several weeks before the race and continuing for a defined recovery period afterward.

Primary Outcome:

-Salivary IgA Concentration The primary outcome is the change in salivary immunoglobulin A (IgA) concentration before and after the competition, assessed at five time points. This measure will reflect mucosal immune function and the potential modulatory effect of daily intake of fermented milk containing Lacticaseibacillus paracasei strain Shirota.

Secondary Outcomes:

* Systemic Immune and Inflammatory Response Blood samples will be analyzed for markers of systemic immune activation and inflammation (e.g., cytokines), collected at five time points to evaluate the broader immunomodulatory effects of the probiotic intervention.
* Upper Airway Symptoms Incidence, severity, and duration of upper airway symptoms (e.g., sore throat, cough, nasal congestion) will be assessed using the Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21). Higher scores indicate more severe symptoms and a greater impact on daily functioning.
* Mood State Mood state changes will be evaluated using the Brunel Mood Scale (BRUMS) across six subscales. Total Mood Disturbance (TMD) scores will reflect the psychological response to training and competition. Higher scores indicate worse mood states.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 25 and 45 years.
* Amateur triathletes with regular endurance training and prior competition experience.
* In good general health, with no history of chronic diseases or conditions affecting immune or inflammatory responses.
* Willing and able to comply with all study procedures, including sample collections and completion of validated questionnaires at five time points.
* Agree to consume a daily dose of fermented milk containing Lacticaseibacillus paracasei strain Shirota (LcS) or placebo from 30 days before until 14 days after the competition.
* No use of probiotics, antibiotics, or immunomodulatory supplements in the 30 days prior to enrollment

Exclusion Criteria:

* Known allergy or intolerance to dairy products, including lactose.
* Use of probiotics or antibiotics within 30 days prior to enrollment.
* Current use of any pharmacological treatment.
* History of chronic rhinopathy.
* Diagnosis of autoimmune disease.
* History of recurrent infections not involving the upper airway.
* Presence of major medical conditions or chronic diseases, including but not limited to respiratory or gastrointestinal disorders.
* Incomplete or missing data necessary for determining eligibility or for study outcomes.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-08-13 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Salivary IgA Concentration | Pre-study: 30 days before the competition (baseline) During study: 24 hours before the competition Post-study: Immediately after the competition, 72 hours post-competition, and 14 days after the competition
  The primary outcome measure is the change in salivary immunoglobulin A (IgA) concentration after daily intake of fermented milk containing Lacticaseibacillus paracasei strain Shirota. Saliva samples will be collected from participants at five time points: 30 days before the competition, 24 hours before, immediately after, 72 hours after, and 14 days post-competition. The concentration of salivary IgA will be measured to assess the impact of probiotic supplementation on immune function.

SECONDARY OUTCOMES:
Immune/Inflammatory Response | Pre-study: 30 days before the competition (baseline) During study: 24 hours before the competition Post-study: Immediately after the competition, 72 hours post-competition, and 14 days after the competition
  The secondary outcome measure is the assessment of systemic immune and inflammatory responses. Blood samples will be collected at five time points: 30 days before the competition, 24 hours before, immediately after, 72 hours after, and 14 days post-competition. These samples will be analyzed for markers of immune activation and inflammation to assess the effects of probiotic supplementation.

OTHER OUTCOMES:
Upper Airway Symptoms | Pre-study: 30 days before the competition (baseline) During study: 24 hours before the competition Post-study: Immediately after the competition, 72 hours post-competition, and 14 days after the competition
  This secondary outcome measures the incidence and duration of upper airway symptoms (e.g., sore throat, cough, nasal congestion) during the study period. Participants will complete the WURSS-21 (Wisconsin Upper Respiratory Symptom Survey-21) questionnaire at five time points: 30 days before, 24 hours before, immediately after, 72 hours after, and 14 days post-competition.
  WURSS-21 Scores Minimum score: 0 (no symptoms) Maximum score: 140 Interpretation: Higher scores indicate more severe symptoms and greater negative impact on daily functioning.
Mood State | Pre-study: 30 days before the competition (baseline) During study: 24 hours before the competition Post-study: Immediately after the competition, 72 hours post-competition, and 14 days after the competition
  The third secondary outcome assesses mood state changes using the Brunel Mood Scale (BRUMS-Profile of Mood States) questionnaire. Participants will complete the questionnaire at five time points: 30 days before the competition, 24 hours before, immediately after, 72 hours after, and 14 days post-competition, to evaluate any effects of probiotic supplementation on mood during the study.
  The BRUMS score consists of 24 items grouped into six subscales: tension, depression, anger, vigor, fatigue, and confusion. Each item is rated on a 5-point scale ranging from 0 ("Not at all") to 4 ("Extremely").
  Minimum score : 0 Maximum score: 96 Interpretation: Higher scores indicate a worse overall mood state.

CONTACTS AND LOCATIONS:
Overall Officials: Jonatas B do Amaral, PHD, Principal Investigator — Federal University of São Paulo; André Luis L Bachi, PHD, Study Chair — Santo Amaro University; Cesar Miguel M dos Santos, PHD, Study Chair — Enau College; Mauro W Vaisberg, PHD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the publication will be shared, after de-identification. This includes salivary IgA concentrations, data on immune and inflammatory markers, upper airway symptoms, and mood state scores (e.g., BRUMS questionnaire).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will be available beginning 6 months after publication of the study results and will remain available for 3 years.
Access Criteria: Researchers who provide a methodologically sound proposal will be able to access the IPD and supporting information. Requests should be directed to the principal investigator by email. A data access agreement will be required prior to sharing.

REFERENCES:
- [Background] Vaisberg M, Paixao V, Almeida EB, Santos JMB, Foster R, Rossi M, Pithon-Curi TC, Gorjao R, Momesso CM, Andrade MS, Araujo JR, Garcia MC, Cohen M, Perez EC, Santos-Dias A, Vieira RP, Bachi ALL. Daily Intake of Fermented Milk Containing Lactobacillus casei Shirota (Lcs) Modulates Systemic and Upper Airways Immune/Inflammatory Responses in Marathon Runners. Nutrients. 2019 Jul 22;11(7):1678. doi: 10.3390/nu11071678. PMID 31336570
- See also: ORL Lab -Official website of the laboratory where the activities will be carried out at the Federal University of Sao Paulo-Brazil — https://ppg.unifesp.br/otorrino/institucional/laboratorio-de-pesquisa-em-otorrinolaringologia-orl-lab
- See also: instagram ORL LAB page — https://www.instagram.com/orl.lab/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT06970964/Prot_SAP_000.pdf